CLINICAL TRIAL: NCT03140124
Title: Enhancing Therapy Process With Movement Strategies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility - unable to recruit therapists to enter the study
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Full Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3889
Record Dates: First submitted 2016-10-07; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Anxiety Disorders; Mood Disorders
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants receive both conditions, with randomized order
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): First session: worry stone, second session: exercise peddler
  Interventions: Behavioral: Exercise; Behavioral: Worry Stone
- Group 2 (Other): First session: exercise peddler, second session: worry stone
  Interventions: Behavioral: Exercise; Behavioral: Worry Stone

INTERVENTIONS:
Behavioral: Exercise — Each participant will be provided with an ActiveLife Trainer to use during visit 2 or 3. The ActiveLife Trainer is a stationary pedaling machine that one can use while seated. It was designed to be used while working and makes very little noise. It is a safe, low-impact physical activity machine with adjustable resistance. The machine communicates via Bluetooth with the Wahoo Fitness app which records activity metrics such as distance cycled. Participants will be provided with a tablet on which the Wahoo Fitness app will track their exercise during the session. The ActiveLife Trainer has been used in numerous research studies (Carr et al., 2014; Botter et al., 2013; Burford et al., 2013; Carr et al., 2013).
Behavioral: Worry Stone — For the worry stone condition, both the participants will rub a stone for the duration of the session. Each participant will be provided with a worry stone to rub during visit 2 or 3. These are small sooth stones that fit in the palm of one's hand.

SUMMARY:
Several studies have noted the benefits of exercise programs in improving both mood and anxiety symptoms. Additionally, single bouts of exercise have been shown to improve mood and anxiety. Business applications report ancillary benefits of exercise as well. For example, individuals spontaneously report better ability to approach stimuli and cope with emotional experiences if doing it while exercising.

The current study aims to investigate exercise during a therapy session as a potential intervention for enhancing therapeutic learning, particularly ability to better cope with emotional topics and experiencing intense emotions. In this study, patient participants will complete a therapy session while using an exercise machine and a separate therapy session while using a worry stone (control). Both patient participants and therapist participants will make ratings of a variety of items, including ability to discuss emotional topics and comfort in experiencing emotions.

Investigators hypothesize that patients will report better ability to discuss emotional topics and more comfort in experiencing emotions following the exercise condition as opposed to the worry stone condition. Investigators also hypothesize that therapist ratings will similarly indicate that patients were better able to discuss emotional topics and experience emotional content during exercise sessions.

DETAILED DESCRIPTION:
The current study aims to investigate exercise during a therapy session as a potential intervention for enhancing therapeutic learning, particularly ability to better cope with emotional topics and experiencing intense emotions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over the age of 18
2. Ability to read and provide informed consent
3. Current patient or therapist at the Center for Anxiety and Related Disorders (CARD)
4. Ability to complete exercise (e.g. no physical injuries)

Exclusion Criteria:

1. Participants considered high risk based on the ACSM risk stratification guidelines (derived from PAR-Q)
2. Participants with current knee, ankle, hip, or foot injuries that could impede exercise on the machine or participants with current hand or wrist injuries that could impede use of the worry stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Session Rating Scale - Patient version (Questions 1 and 2) | Change throughout 50-minute therapy session.
  Patients will be asked questions on a 1 to 5 Likert scale examining degree to which they discussed emotional topics during session (Question 1) and the degree to which they felt comfortable discussing emotional topics during session (Question 2).
Session Rating Scale - Therapist version (Questions 1 and 2) | Change throughout 50-minute therapy session.
  Therapists will be asked questions on a 1 to 5 Likert scale examining degree to which they felt their patients discussed emotional topics during session (Question 1) and the degree to which they felt their patients were comfortable discussing emotional topics during session (Question 2).

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule - Patient | Change throughout 50-minute therapy session.
  State Version (PANAS; Watson, Clark, & Tellegen, 1988). The PANAS was developed as a brief measure of affect and yields the factors of Positive Affectivity and Negative Affectivity.
Positive and Negative Affect Schedule - Therapist | Change throughout 50-minute therapy session.
  State Version (PANAS; Watson, Clark, & Tellegen, 1988). The PANAS was developed as a brief measure of affect and yields the factors of Positive Affectivity and Negative Affectivity.
Affect Grid - Patient | Change throughout 50-minute therapy session.
  A single item scale used to quickly assess affect along the dimensions of pleasure-displeasure and arousal-sleepiness
Affect Grid - Therapist | Change throughout 50-minute therapy session.
  A single item scale used to quickly assess affect along the dimensions of pleasure-displeasure and arousal-sleepiness
Credibility-Expectations Questionnaire - Patient | Change throughout 50-minute therapy session.
  The CEQ is a 6-item self-report questionnaire, which assesses treatment rationale and expectancy. The scale has been used across a number of treatment trials. This questionnaire will be slightly modified to measure satisfaction with the worry stone and exercise machine conditions and will be administered at the beginning of each visit.
Credibility-Expectations Questionnaire - Therapist | Change throughout 50-minute therapy session.
  The CEQ is a 6-item self-report questionnaire, which assesses treatment rationale and expectancy. The scale has been used across a number of treatment trials. This questionnaire will be slightly modified to measure satisfaction with the worry stone and exercise machine conditions and will be administered at the beginning of each visit.
Session Rating Scales (Questions 3-7) - Patient | Change throughout 50-minute therapy session.
  Participants will be asked questions on a 1 to 5 Likert scale related to involvement of the intervention in ability to discuss emotional topics and comfort in using the intervention device.
Session Rating Scales (Questions 3-7) - Therapist | Change throughout 50-minute therapy session.
  Participants will be asked questions on a 1 to 5 Likert scale related to involvement of the intervention in ability to discuss emotional topics and comfort in using the intervention device.
Qualitative Feedback - Therapist | Change throughout 50-minute therapy session.
  Therapists will be given the option to write briefly about their thoughts of the impact of the movement strategies on their therapy sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No